CLINICAL TRIAL: NCT06390397
Title: Brighter Bites & University of Texas Physicians Produce Rx Extension: Evaluating the Effectiveness of a Prospective Clinical Nutrition Study With Produce Prescriptions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Brighter Bites and Humana Foundation (Unknown)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-24-0129
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Produce prescription program (Experimental)
  Interventions: Other: Produce prescription program; Other: Standard of care
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Produce prescription program — Boxes of fresh fruit and vegetables (F&V), each containing approximately 50 servings of F&V, will be assembled by Brighter Bites at school sites using donated produce and delivered to houses using DoorDash. F&V boxes will be distributed to families every 2 weeks over 32 weeks. Participants will also receive nutrition education using the Brighter Bites app which includes recipes for a variety of meal types or produce types, all of which are searchable. Recipes include the average cost to prepare, the number of servings, and the calories for the recipe. The Brighter Bites app also includes healthy living "Brighter Choices" suggestions such as tips for how to store different types of foods, gardening tips, and tips to pack a healthy lunchbox. In addition to the Brighter Bites app, trained staff will facilitate virtual nutrition education for patient families.
  Arms: Produce prescription program
Other: Standard of care — Standard of care includes routine lab work collection and weight and diet counseling for overweight or obese children. Additionally, referrals placed to community resources for those identified with Social Determinants of Health(SDOH) needs.

SUMMARY:
The purpose of this study is to clinically evaluate the effectiveness of an at-home delivery produce prescription in improving weight status and obesity-related health outcomes and to examine the impacts of the program on child dietary behavioral outcomes (child fruit and vegetable intake, junk food consumption, and eating at any type of restaurant), and parent feeding practices (preparing foods from scratch, use of nutrition facts labels to make purchasing decisions, and eating meals with their referent child).

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at University of Texas Physicians Greens Clinic or University of Texas Physicians Pediatric Primary Care in Houston, Texas
* BMI>85th percentile
* reside within a 10-mile radius of a Brighter Bites school
* Medicaid recipients or low-income uninsured
* parents must be able to read and write in English or Spanish to complete surveys

Exclusion Criteria:

* currently participating in Brighter Bites
* a family member/sibling currently participating in Brighter Bites
* child is currently attending a school that offers Brighter Bites

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | baseline , post intervention (32 weeks after baseline)
Change in systolic blood pressure | baseline , post intervention (32 weeks after baseline)
Change in diastolic blood pressure | baseline , post intervention (32 weeks after baseline)
Change in level of hemoglobin A1c in milligrams per deciliter (mg/dL) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in level of Aspartate transaminase (AST) in units per liter (U/L) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in level of Alanine transaminase (ALT) in units per liter (U/L) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in level of low-density lipoprotein(LDL) in milligrams per deciliter (mg/dl) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in levels of high-density lipoprotein(HDL) in milligrams per deciliter (mg/dl) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in levels of total cholesterol in milligrams per deciliter (mg/dl) as assessed by blood work | baseline , post intervention (32 weeks after baseline)
Change in levels of triglycerides in milligrams per deciliter (mg/dl) as assessed by blood work | baseline , post intervention (32 weeks after baseline)

SECONDARY OUTCOMES:
Change in amount of fruit and vegetable intake | baseline , post intervention (32 weeks after baseline)
Change in amount of junk food consumed | baseline , post intervention (32 weeks after baseline)
Change in number of times subject eats out at restaurants | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has cooked food from scratch | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has used nutrition facts labels to make purchasing decisions | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has eaten meals with their referent child | baseline , post intervention (32 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No